CLINICAL TRIAL: NCT04152252
Title: Cardio-Pulmonary-Resuscitation Quality in Out-of-Hospital Cardiac Arrest - Effect of Real-time Feedback and Post-event Debriefing
Brief Title: CPR Quality and Use of Feedback for OHCA
Status: Completed | Type: Observational
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: TrygFonden, Denmark (Industry); St George's, University of London (Other); Kingston University (Other)
Responsible Party: Principal Investigator, Rasmus Meyer Lyngby, Paramedic (BSc.), Emergency Medical Services, Capital Region, Denmark
Other Study IDs: F-35103-02
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: OHCA; Feedback; CPR quality
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Baseline: No CPR feedback during CPR
- Real-time feedback: Real-time feedback on chest compression depth, chest compression rate and recoil available to EMS while performing CPR. Feedback is delivered as visual text, numeric and graphical presentations on the defibrillator with audio tones for rate.
  Interventions: Other: Real time feedback
- Post-event debriefing: Structured oral post-event debriefing based on objective performance data from the resuscitation attempt. The debriefing is conducted as hot/immediate self-directed debriefing session with a maximum length of 10 minutes.
  Interventions: Other: Real time feedback; Behavioral: Post-event debriefing

INTERVENTIONS:
Other: Real time feedback — Real-time feedback on chest compression depth, chest compression rate and recoil available to EMS while performing CPR. Feedback is delivered as visual text, numeric and graphical presentations on the defibrillator with audio tones for rate.
  Groups: Post-event debriefing; Real-time feedback
Behavioral: Post-event debriefing — Structured oral post-event debriefing based on objective performance data from the resuscitation attempt. The debriefing is conducted as hot/immediate self-directed debriefing session with a maximum length of 10 minutes.
  Groups: Post-event debriefing

SUMMARY:
The purpose of this study is to investigate the quality of cardio-pulmonary resuscitation(CPR) delivered by EMS professionals and whether this quality can be improved by implementing real-time feedback during the event and an oral post-event debriefing procedure based on the actual event performance data.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether CPR quality can be improved by implementing real-time feedback and immediate oral structured post-event debriefing in out-of-hospital cardiac arrest (OHCA).

The objectives of this study is to assess the current quality of CPR delivered by emergency medical services (EMS) during OHCA events in the Capital Region of Denmark. Furthermore, to investigate if CPR quality can be improved by applying real-time feedback during OHCA resuscitation attempts and to investigate if structured oral post-event debriefing delivered immediately after a resuscitation attempt and based on data from the defibrillator can further improve CPR quality

The hypothesis of this study is that adding real-time and post event feedback can improve the compression rate, compression depth, overall CPR hands-on time (CPR fraction), and recoil with at least 15% in total for both interventions.

Using a prospective study design data is retrieved from the standard defibrillator (ZOLL X series) through ZOLL RescueNet® Case Review (software for post-event review, analysis, and debriefing) from ZOLL Medical Corporation, Massachusetts, United States of America.

The study consists of three consecutive phases. Phase one with no feedback / debriefing available for EMS. Phase two with real-time feedback during the event and phase three which adds post-event debriefing to real-time feedback. We expect to be able to include at least 500 cases in each phase.

ELIGIBILITY:
Inclusion Criteria:

OHCA

Exclusion Criteria:

No use of EMS defibrillator attached to patient during resuscitation attempt Patients < 18 years of age OHCA without involvement of the physician manned vehicle Patients who are subject to mechanical CPR from the time of device attachment Traumatic OHCA

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients in OHCA in the Capital Region of Denmark who receive CPR by or under supervision of EMS professionals with the standard EMS defibrillator attached.
Sampling Method: Non-Probability Sample
Enrollment: 2989 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Chest compression depth | During cardiopulmonary resuscitation performed by emergency medical services, up to 4 hours
  Chest compression depth is defined as the maximum posterior deflection of the sternum prior to chest recoil. Measured in centimeters and as percentage of compressions within the recommended 5 to 6 cm

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | During cardiopulmonary resuscitation performed by emergency medical services, up to 4 hours
  The return of a spontaneous pulse prior to handover at hospital measured as events
Sustained return of spontaneous circulation (ROSC) | During cardiopulmonary resuscitation performed by emergency medical services, up to 4 hours
  The return of a spontaneous pulse at hospital handover measured as events
30- day survival | 30 days from event
  Patient alive at day 30 from event
Chest compression rate | During cardiopulmonary resuscitation performed by emergency medical services, up to 4 hours
  Chest compression rate is defined as the frequency of chest compressions during compression series. Measured in number compressions per minute (cpm) and percentage of delivered compressions within the recommended rate of 100-120 cpm
Chest compression fraction | During cardiopulmonary resuscitation performed by emergency medical services, up to 4 hours
  Chest compression fraction is defined as the time with chest compressions starting from the first therapeutic event to the end of the episode. An episode is the time without presence of a spontaneous patient pulse. Measured in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Lyngby, BSc, Principal Investigator — Emergency Medical Services, Capital Region, Denmark
Locations (1):
- Copenhagen EMS, Ballerup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No
Danish legislation do not allow for sharing of individual patient data without patient consent

REFERENCES:
- [Derived] Lyngby RM, Quinn T, Oelrich RM, Nikoletou D, Gregers MCT, Kjolbye JS, Ersboll AK, Folke F. Association of Real-Time Feedback and Cardiopulmonary-Resuscitation Quality Delivered by Ambulance Personnel for Out-of-Hospital Cardiac Arrest. J Am Heart Assoc. 2023 Oct 17;12(20):e029457. doi: 10.1161/JAHA.123.029457. Epub 2023 Oct 13. PMID 37830329